CLINICAL TRIAL: NCT01306123
Title: An Open, Randomized, Single-dose, Two-way Crossover Study to Characterize the Pharmacokinetic Properties of Cyanocobalamin When Administered as an Intranasal Spray and an Intramuscular Injection to Healthy Volunteers
Brief Title: Characterization of Cyanocobalamin in Healthy Voluteers After Intranasal and Intramuscual Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NSB09/17
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Focus: Bioavailability
Keywords: bioavailability; pharmacokinetics; cyanocobalamin; intranasal; intramuscular
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nascobal nasal spray (cyanocobalamin USP) (Experimental): One single administration of intranasal cyanocobalamin (initially)
  Interventions: Drug: Nascobal nasal spray (cyanocobalamin, USP)
- Vitamin B12-ratiopharm N, injection solution (Active Comparator): One single injection of IM cyanocobalamin (initially)
  Interventions: Drug: Vitamin B12-ratiopharm N, injection solution

INTERVENTIONS:
Drug: Nascobal nasal spray (cyanocobalamin, USP) — Single intranasal administration
  Arms: Nascobal nasal spray (cyanocobalamin USP)
Drug: Vitamin B12-ratiopharm N, injection solution — One single intramuscular administration
  Arms: Vitamin B12-ratiopharm N, injection solution

SUMMARY:
The main purpose of this study is to assess the relative bioavailability of Nascobal Nasal Spray as compared to an IM injection of cyanocobalamin (European reference product).

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose, two-way crossover study. The study consists of a screening visit, two 4-days confinement periods and a follow-up telephone call. The two confinement periods will be separated by a washout period of at least 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female and male voluteers
* 18-40 years of age
* BMI between 18.5 and 30.0 kg/m2

Exclusion Criteria:

* Females who are pregnant or lactating
* History of clinically significant metabolic, hepatic, renal, haematological, pulmondary, cardiovascular, gastrointestinal, urological, neurological or phychiatric disorders
* Serum vitamin B12 <=250 pmol/L or MMA >=0.40 umol/L
* Evidence of significant intranasal pathology
* Nasal congestion, allergic rhinitis or upper respiratory tract infection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability | 0-72 hours
  Relative bioavailability (Frel) based on the area under the serum concentration-time curve during 72 hours (AUC0-72h) for the test and reference products.

SECONDARY OUTCOMES:
Additional PK characteristics | 0-72h
  Maximum serum concentration (Cmax), time of Cmax (tmax) and AUC0-24h.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Al-Tawil, MD, PhD, Principal Investigator — Karolinska Trial Alliance
Locations (1):
- Karolinska Trial Alliance, Karolinska University Hospital, Huddinge, Stockholm, Stockholm County, Sweden